CLINICAL TRIAL: NCT00468078
Title: The Single Center, Phase III Clinical Trial to Evaluate the Efficacy and the Safety of [18F]FPCIT Positron Emission Tomography in Parkinson's Disease and Essential Tremor Patients
Brief Title: Efficacy and Safety of F-18 FPCIT PET in Parkinson's Disease and Essential Tremor Patients
Acronym: FPCIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jae Seung Kim, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: FPCITKR001
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Essential tremor; F-18 FPCIT; PET
MeSH Terms: conditions — Parkinson Disease; Essential Tremor | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Parkinson's disease
  Interventions: Procedure: PET/CT; Drug: F-18 FPCIT
- B (Active Comparator): ET+Normal
  Interventions: Procedure: PET/CT; Drug: F-18 FPCIT

INTERVENTIONS:
Procedure: PET/CT — 10min acquisition, 90min after injection of F-18 FPCIT
  Other Names: Positron Emission Tomography
Drug: F-18 FPCIT — 5mCi, intravenous injection

SUMMARY:
The purpose of this study is to determine whether F-18 FPCIT is effective and safe radiopharmaceutical for the objective diagnosis of Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a common neurodegenerative disorder with loss of dopaminergic terminals in the striatum. Essential tremor is one of the conditions most commonly misdiagnosed as parkinsonism, and early clinical differentiation between these conditions can be difficult. F-18 FPCIT is a promising radiopharmaceutical for PET imaging to assess the dopamine transporter in the striatum.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's disease

* Male or female with age over 40 years
* Clinical diagnosis of Parkinson's disease
* Ability to give informed consent

Essential tremor

* Male or female with age over 40 years
* Clinical diagnosis of Essential tremor
* Ability to give informed consent

Healthy volunteers

* Male or female with age over 40 years
* No any symptoms or sign suggesting Parkinson's disease or essential tremor
* Ability to give informed consent

Exclusion Criteria:

Parkinson's disease and essential tremor

* Current pregnancy and breast feeding
* Current or past medical history of cardiac and neuropsychiatric disease
* Clinical evidence of dementia
* Inability to hold antiparkinsonian medication
* History of surgical therapy for tremor
* Severe or unstable medical or psychiatric condition
* Medication affecting CNS in last 6 months(e.g. CNS stimulants, sympathomimetics)
* Prior participation in other research protocol within 30 days

Healthy volunteers

* Current pregnancy and breast feeding
* Current or past medical history of cardiac and neuropsychiatric disease
* Severe or unstable medical or psychiatric condition
* Drug abuse or medication affecting CNS (e.g. CNS stimulants, sympathomimetics) within 6 months
* Prior participation in other research protocol within 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
diagnostic sensitivity and specificity, and acute complication | 1 month

SECONDARY OUTCOMES:
correlation of specific striatal uptake to non specific uptake ratio of F-18 FPCIT and clinical sererity (H&Y stage) | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jae Seung Kim, MD, Principal Investigator — Department of Nuclear Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Kazumata K, Dhawan V, Chaly T, Antonini A, Margouleff C, Belakhlef A, Neumeyer J, Eidelberg D. Dopamine transporter imaging with fluorine-18-FPCIT and PET. J Nucl Med. 1998 Sep;39(9):1521-30. PMID 9744335